CLINICAL TRIAL: NCT06437808
Title: Optimizing Football Training at Multan Sports Complex: Integrating Portable Force Plates for Advanced Performance Analysis
Brief Title: Optimizing Football Training: Integrating Portable Force Plates for Advanced Performance Analysis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSRSW/Batch-Fall22/716
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Injury;Sports
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training with Portable Force Plates Integration (Experimental)
  Interventions: Combination Product: Training with Portable Force Plates Integration
- Standard Training (Other)
  Interventions: Other: Standard Training

INTERVENTIONS:
Combination Product: Training with Portable Force Plates Integration — This group will undergo football training sessions that incorporate the use of portable force plates. These devices will measure ground reaction forces and provide real-time data on players' movements, balance, and pressure points. The data collected will be used to create personalized training programs aimed at optimizing performance and reducing the risk of injuries.
  Arms: Training with Portable Force Plates Integration
Other: Standard Training — This group will continue with the existing football training regimen without the use of portable force plates. Training will follow the traditional methods used at the Multan Sports Complex, focusing on physical conditioning, technical skills, and tactical awareness without the advanced biomechanical analysis provided by the force plates.
  Arms: Standard Training

SUMMARY:
Optimizing Football Training at Multan Sports Complex: Integrating Portable Force Plates for Advanced Performance Analysis," aims to enhance football training through innovative technology. Under the supervision of Dr. Junaid Gondal, this MS Rehabilitation Science project explores the use of portable force plates to provide real-time data on players' biomechanics, enabling personalized training programs that improve performance and reduce injury risks.

DETAILED DESCRIPTION:
The research adopts a randomized control trial design, involving 30 male football players aged 18-35. Participants are divided into intervention and control groups, with the former using portable force plates during training. Data analysis will be conducted using IBM SPSS. This study underscores the significance of advanced performance analysis in football training, advocating for the integration of cutting-edge technology to refine training methods and enhance athletic performance at the Multan Sports Complex.

ELIGIBILITY:
Inclusion Criteria:

* Male football players at Multan Sports Complex
* aged 18-35
* willing to consent.

Exclusion Criteria:

* Female players
* unregistered players
* those with unstable medical conditions.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-29 (Estimated)

PRIMARY OUTCOMES:
RPE Scale | 12 Months
  Rate of perceived exertion (RPE) is used to measure how hard your body works during physical activity. It runs from 0 - 10, using numbers to rate how much effort an activity takes

CONTACTS AND LOCATIONS:
Locations (1):
- Multan Sports Complex, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No